## NCT02714153

Bridge Occlusion Balloon in Lead Extraction Procedure SAP

8/2020

Baseline characteristics were reported as mean and standard deviation for continuous data and frequencies and percentages for categorical data. Serial procedural hemodynamic measures were assessed with repeated measures analysis of variance. Statistical significance was set at p<0.05 for all comparisons using two-way ANOVA.